CLINICAL TRIAL: NCT03297164
Title: One Year Incidence Rate of Heart Failure After Acute Myocardial Infarction With Optimal Treatment-A Prospective,Multicenter,Cohort Study
Brief Title: Incidence Rate of Heart Failure After Acute Myocardial Infarction With Optimal Treatment
Status: Completed | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, director, Harbin Medical University
Other Study IDs: 2016YFC1301101
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: acute myocardial infarction; heart failure; optimized treatment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- optimized group: the patients in this group have been given the suggestive treatment from guideline.
- un-optimized group: the patients in this group have not been given the suggestive treatment from guideline.

SUMMARY:
The main purpose of this study is to build a multi-center, prospective and regionally representative acute myocardial infarction(AMI) cohort，and build a study platform for heart failure caused by AMI; To explore the 1 year incidence rate of heart failure after AMI given the optimized treatment and the treatment model affecting the incidence rate of heart failure, and finally to reduce the incidence rate of heart failure by 5%.

DETAILED DESCRIPTION:
the study aim to enroll 12000 acute myocardial infartion (AMI) patients, including ST-segment elevation myocardial infarction (STEMI) and non ST-segment elevation myocardial infarction (NSETMI), Patients were divided into two groups(optimized group and un-optimized group) according to treatment models they accepted in 20 reginally representative hosptials of China. whether optimizaed or not is judged by 4 four aspects,including emergency treatment procedure, pre-infusion medication, reperfusion strategy selection, and early rehabilitation after reperfusion.Patients were followed at 1 month, 6 months and 12 months. The physical condition and clinical events(heart failure, death, re-infarction, revascularization, apoplexy, malignant arrhythmias, bleeding events, other adverse events)were collected at follow up.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* diagnosed acute myocardial infarction
* signed the informed consent form

Exclusion Criteria:

* AMI is caused by surgery, trauma, gastrointestinal bleeding or complications of PCI;
* AMI occurred in patients who have been hospitalized for other reasons;
* patients with previous history of chronic heart failure;
* researchers judging that patient's compliance was poor and could not complete the study according to the requirements.
* life expectancy is less than 12 months;
* heart transplant patients;
* patients with tumors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute myocadial infarction
Sampling Method: Non-Probability Sample
Enrollment: 12043 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
incidence rate of heart failure | 12th month after diacharge
  incidence rate of heart failure of acute myocardial infarction at 12th month

SECONDARY OUTCOMES:
MACCE rate | 12th month after diacharge
  the major adverse cardiac celebral events including death,reinfarction,
bleeding rate | 12th month after diacharge
  the incidence rate of bleeding
severe adverse drug reactions | 12th month after diacharge
  severe adverse drug reactions at 12th month

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beijing An Zhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Univerisity People'Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guangdong general hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Guangxi medical university, Nanning, Guangxi
  - Second hospital of hebei medical university, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The first affiliated hospital of Zhengzhou medical university, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - the second affiliated hospital of Dalian medical university, Dalian, Liaoning
  - Shenyang military district general hospital of the people's liberation army, Shenyang, Liaoning
  - The first affiliated hospital of military medical university, Xi’an, Shanxi
  - Third Military Medical University, Chongqing, Sichuan
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Li Z, Yang G, Fang C, Yin Y, Zheng Z, Wang H, Fang S, Dai J, Wang S, Yang S, Yu B. Pseudo-targeted metabolic profile differences between emergency patients with type 1 and type 2 myocardial infarction diagnosed by optical coherence tomography. Clin Chim Acta. 2024 Feb 1;554:117745. doi: 10.1016/j.cca.2023.117745. Epub 2024 Jan 6. PMID 38185283
- [Derived] Lang X, Zhao B, Fang S, Li L, Li Z, Wu N, Zhang Y, Xing L, Li Y, Zhang Y. Higher Peripheral Thyroid Sensitivity Is Linked to a Lower Risk of Heart Failure After Acute Myocardial Infarction. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2950-2960. doi: 10.1210/clinem/dgad240. PMID 37104944
- [Derived] Zeng M, Zhao C, Bao X, Liu M, He L, Xu Y, Meng W, Qin Y, Weng Z, Yi B, Zhang D, Wang S, Luo X, Lv Y, Chen X, Sun Q, Feng X, Gao Z, Sun Y, Demuyakor A, Li J, Hu S, Guagliumi G, Mintz GS, Jia H, Yu B. Clinical Characteristics and Prognosis of MINOCA Caused by Atherosclerotic and Nonatherosclerotic Mechanisms Assessed by OCT. JACC Cardiovasc Imaging. 2023 Apr;16(4):521-532. doi: 10.1016/j.jcmg.2022.10.023. Epub 2022 Dec 14. PMID 36648054
- [Derived] Li L, Zhang X, Wang Y, Yu X, Jia H, Hou J, Li C, Zhang W, Yang W, Liu B, Lu L, Tan N, Yu B, Li K. A Novel Risk Score to Predict In-Hospital Mortality in Patients With Acute Myocardial Infarction: Results From a Prospective Observational Cohort. Front Cardiovasc Med. 2022 Apr 7;9:840485. doi: 10.3389/fcvm.2022.840485. eCollection 2022. PMID 35463775